

# UNIVERSITY OF CALIFORNIA, SAN FRANCISCO CONSENT TO PARTICIPATE IN A RESEARCH STUDY

# CC#122011: A PHASE II STUDY OF RADIATION THERAPY AND VISMODEGIB, FOR THE TREATMENT OF LOCALLY ADVANCED BASAL CELL CARCINOMA OF THE HEAD AND NECK

This is a clinical trial, a type of research study. Your study doctors, Sue S. Yom, M.D. and Roy Grekin, M.D. and their associates from the University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center will explain the clinical trial to you.

Clinical trials include only people who choose to take part. Please take your time to make your decision about participating. You may discuss your decision with your family and friends and with your health care team. If you have any questions, you may ask your study doctor.

You are being asked to take part in this study because you have a locally advanced basal cell carcinoma, a type of skin cancer.

#### WHY IS THIS STUDY BEING DONE?

Chemotherapy, radiation therapy, and surgery are standard treatments for basal cell carcinoma at most institutions. The purpose of this study is to determine whether adding vismodegib to radiation (chemoradiotherapy) is safe and tolerable. The purpose of this study is to assess the safety and tolerability of combined radiation therapy and vismodegib. This combination may increase the chances of the tumors being destroyed or unable to spread to other parts of the body in people with locally advanced basal cell carcinoma of the head and neck.

Vismodegib has been approved by the US Food and Drug Administration (FDA) for the treatment of basal cell carcinoma. It may delay the growth of tumor cells. In previous studies of vismodegib in humans with basal cell carcinoma, vismodegib has shown an anti-tumor effect.

The combination of vismodegib and radiation therpay is considered experimental; that means this combination has not been approved by the FDA.

Genentech, a member of the Roche group, is providing funding to UCSF to conduct the study. Genenetch, the manufacturer of study drug, will also provide the study drug at no cost to study participants.

## HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 24 people may participate in the study. About 20 people will take part in this study at UCSF, San Francisco General Hospital, and the San Francisco VA Medical Center.

#### WHAT WILL HAPPEN IF I TAKE PART IN THIS RESEARCH STUDY?

### Study treatment

Vismodegib will be taken daily, once a day on an empty stomach either 1 hour before or 2 hours after meals for 12 weeks, then for 1-14. days as required until the start of radiation therapy. You should take the study drug at approximately the same time each day. You will be given a supply of vismodegib on Week 1, Day 1 to last until your next study visit. You will be asked to keep a record of each dose of vismodegib you take. After 12 weeks, you will be evaluated again to make sure you are still eligible to participate in the study. If you are eligible to continue, you will continue taking vismodeib daily as before for another 7 weeks while you receive radiation therapy.

Radiation therapy will be started after you have finished taking vismodegib for 12 weeks. You will receive radiation once a day, Monday through Friday, for 7 weeks. Each radiation treatment may take up to 30 minutes.

# Before you begin the main part of the study...

You will need to have the following exams, tests or procedures to find out if you can be in the main part of the study. These exams, tests or procedures are part of regular cancer care and may be done even if you do not join the study. You will also have some procedures that are only being done because you are in the study. These are called research procedures and are noted in the list of procedures below. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor. The total time needed to complete all screening tests and procedures is approximately 8 hours.

# Within 28 days of beginning study treatment:

- Complete history
- Tumor assessment by CT (Computed Tomography) scan or MRI (Magnetic Resonance Imaging) scan
  - o A CT scan uses special x-ray equipment to make detailed pictures of body tissues and organs. For the CT scan, you may be given a "contrast material" (a special dye that makes it easier for doctors to see different tissues in your body). The contrast material may be given orally, intravenously, or rectally (less likely). Oral contrast material is given to you to drink and is used to help outline the stomach and intestines. Intravenous (IV) contrast material is given to you by injecting the contrast material into a line which is attached to a needle in your arm, and is used to get clearer pictures of your body cavity. A rectal contrast fills up the loops of your lower bowel so the doctors can see your tumor better. After you have been given the contrast material (either by mouth, by vein, or rectum), you will lie flat on a table that will move you into the CT scan machine. You will be asked to lie still and may be asked to hold your breath for a few seconds. The CT scan is done in the radiology department and takes about half an hour.
  - An MRI scan takes an image of your skull or body to observe the location and size of your tumor. For the MRI scan, you may be given a "contrast material" (a special dye that makes it easier for doctors to see different tissues in your body). Gadolinium is contrast material that causes some tumors to appear much brighter than normal tissue on MRI scans (these tumors may not be visible without gadolinium). The contrast material may be given to you in your arm through an intravenous catheter (a tiny tube inserted into a vein). You will then lie down on a narrow bed which will be placed in a tunnel that is 6 feet long by 22 inches wide and open at each end. You will lie there quietly for about one hour, during which time you will hear a loud machine-like noise. The MRI scan is done in the radiology department and takes approximately an hour and a half to complete.
- Chest X-ray or CT (Computed Tomography) chest
  - A chest x-ray will be done that will allow doctors to look at the heart, lungs, and bones. This will take approximately 15-30 minutes to complete.
  - CT Chest as described above but focused on the chest area
- If you have visible tumors on your body, you will also have a tumor biopsy. The biopsy can be done up to 360 days prior to starting study treatment. While participating in the study, if your study doctor suspects that your disease is progressing, you will have another tumor biopsy for confirmation.

Tumor biopsy - A doctor will remove a piece of your tumor tissue if it can be obtained. This is called a biopsy. Usually, this biopsy involves the use of a small needle which is directed into your tumor site with the guidance of an imaging machine such as a CT scan or a Doppler ultrasound, if necessary. This procedure takes about 30 minutes. You will sign a separate consent form for this procedure.

# Within 14 days of beginning study treatment

- Physical exam, including height, weight, and baseline conditions
- Review of the medications you are taking
- Evaluation of adverse events
- Concomitant medications
- Assessment of your ability to perform everyday tasks
- Vital signs (heart rate, body temperature, respiratory rate, blood pressure)
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age. This procedure will be performed 7 days before receiving the study drug.
- Urine test
- If you have visible tumors on your body, your study doctor will take measurements of the tumors

The following tests may be recommended by your study doctor:

- PET/CT(Positron Emission Tomography /Computed Tomography)
  - A PET/CT scan can show how the organs and cells work in your body and is done to show activity of the cells in your tumor. For this procedure, an IV is started in the hand. A small amount of radioactive chemical (glucose) is injected into the blood stream. Once the glucose is injected, you will be asked to wait for about an hour to allow for glucose to distribute in the body. Then you will be asked to lie down on a table and the body is scanned. The total time one will spend at the clinic is about 2-3 hours.
- o Brain MRI see description above
- o Fine Needle Biopsy to confirm if regional nodes are involved regional nodes
  - If you agree to have a tissue biopsy of a lymph node, the skin over the lymph node will first be cleaned with an iodine solution. The skin will then be numbed with lidocaine, after which a needle (slightly larger than the ones used for blood draws) will be inserted one or more times to obtain a tiny amount of tissue within the needle. The needle puncture site should not require more than light pressure for a few minutes to stop the bleeding. You may have some soreness and occasionally a bruise may result. This procedure will take about 30 minutes.
- o For patients with head and neck cancers where radiation will be delivered to the mouth or salivary glands, dental evaluation is strongly recommended

The following procedure will be done for research:

• If you have visible tumors on your body, photographs will be taken of the lesion. This is important because basal cell carcinoma can spread to other areas of your skin. Your face will not be in the photographs unless the basal cell carcinoma affects parts of your face, in which case your eyes will be covered. Your doctor will be particularly careful to respect your confidentiality in this part of the trial. This will take about 5-10 minutes.

Skindex-16 survey

# During the main part of the study...

If the exams, tests and procedures show that you can be in the main part of the study, and you choose to take part, then you will need the following tests and procedures. Each visit will take less than 1 hour.

You will start taking vismodegib on week 1, day 1 and continue to take it once a day. You will be given your supply once you have completed all of the screening tests.

# Week 5 and 9 (Induction Phase)

- Physical examination including weight
- Vital signs
- Performance status
- Evaluation of adverse events
- Concomitant medications
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age week 5

The following procedure will be done for research:

Urine or blood pregnancy test - if a woman of childbearing age – weeks 9 only

# Week 13-14 (End of Induction Phase)

Within 14 days after you have completed 12 weeks of taking vismodegib, you will be reevaluated to make sure you are still eligible to participate in the study. You will have the following procedures. The visit will take about 2-3 hours.

- Physical examination including weight
- Vital signs
- Performance status
- Evaluation of adverse events
- Concomitant medications
- Skindex-16 survey study test
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age
- Imaging (CT or MRI) of head and neck for tumor assessment
- Imaging (CT) of chest or chest x-ray if clinically indicated
- If you have visible tumors on your body, your study doctor will take measurements of the tumors
- You will continue to taking vismodegib once a day

The following procedures will be done for research:

- Skindex-16 survey
- If you have visible tumors on your body, photographs will be taken of the lesion.

# **Week 15-21 (Combination Therapy)**

- Limited physical exam
- Evaluation of adverse events
- Concomitant medications
- You will receive radiation once a day, Monday through Friday, for 7 weeks. Each radiation treatment may take up to 30 minutes.
- You will continue taking vismodegib once a day

## Week 18 only:

- Urine test
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age (this is a research test)

# When you are finished receiving vismodegib and radiation therapy...

## End of treatment visit

You will have an End of treatment visit within 8 -12 weeks of the last dose of vismodegib and radiation therapy. The visit will take about 4 hour(s) and the following tests and procedures will occur:

- Physical examination including weight
- Vital signs
- Performance status
- Evaluation of adverse events
- Concomitant medications
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age
- Imaging (CT or MRI) of head and neck for tumor assessment
- Imaging (CT) of chest or chest x-ray if clinically indicated
- If you have visible tumors on your body, your study doctor will take measurements of the tumors

The following procedures will be done for research:

• Skindex-16 survey
If you have visible tumors on your body, photographs will be taken of the lesion.

## Follow-Up Visits

The study team will ask you to return to the clinic at 3, 6, and 12 months (+/- 2 weeks) after the end of study visit. Each visit will take about 4 hours. You will have the following procedures.

- Physical examination including weight
- Vital signs
- Performance Status

- Evaluation of adverse events
- Concomitant medications
- Blood (about 2 teaspoons) will be drawn for routine safety tests
- Urine or blood pregnancy test if a woman of childbearing age 3 and 6 month visits only
- Imaging (CT or MRI) of head and neck for tumor assessment only at 6 month visit
- Imaging (CT) of chest or chest x-ray if clinically indicated, only at 6 month visit
- If you have visible tumors on your body, your study doctor will take measurements of the tumors

The following procedures will be done for research:

- Skindex-16 survey
- If you have visible tumors on your body, photographs will be taken of the lesion.

After 1 year, the study team would like to keep track of your medical condition for 1 more year. We would like to do this by calling or reviewing your medical record every 3 months to see how you are doing. Keeping in touch with you and checking on your condition helps us look at the long-term effects of the study.

**Study location:** All study procedures will be done at the Helen Diller Family Comprehensive Cancer Center at UCSF or San Francisco General Hospital.

#### HOW LONG WILL I BE IN THE STUDY?

You will receive vismodegib for up to 21 weeks (approximately 5.5 months) and radiation therapy for seven weeks during week 15-21 of vismodegib therapy. You will continue to receive study treatment as long as your disease does not progress or you do not have severe side effects, you experience any bad side effects, you decide to withdraw your consent to participate in this study, or the study is closed.

After you are finished taking the treatment, the study doctor will ask you to visit the office for follow-up exams within 8-12 weeks and then 3, 6, and 12 months (+/- 2 weeks) later. After one year, to follow up on your health status, we would like to call or review your medical records every 3 months for up to 1 more year to see how you are doing.

Keeping in touch with you and checking on your condition helps us look at the long-term effects of the study. Even if your disease has progressed, the study team would like to continue to monitor your health outcomes. Please let the study doctor know if you do not want to participate in this portion of the study.

## **CAN I STOP BEING IN THE STUDY?**

Yes. You can decide to stop at any time. Tell the study doctor if you are thinking about stopping or decide to stop, they will tell you how to stop safely.

It is important to tell the study doctor if you are thinking about stopping so any risks from the vismodegib and radiation therapy can be checked by your doctor. Another reason to tell your doctor that you are thinking about stopping is to talk about what follow-up care and testing could be most helpful for your cancer treatment.

The study doctor may stop you from taking part in this study at any time if they believe it is in your best interest, if you do not follow the study rules, or if the study is stopped.

# WHAT SIDE EFFECTS OR RISKS CAN I EXPECT FROM BEING IN THE STUDY?

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. Side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking vismodegib and radiation. In some cases, side effects can be serious, long lasting, or may never go away. There also is a risk of death.

Handling vismodegib and having contact with any urine, feces or vomit from patients receiving vismodegib may pose some risk to you and your caregivers. To avoid exposure to vismodegib and any associated risks, you and your family members/caregivers will be educated by a member of the study team on how to safely handle, properly dispose of, and clean products that may be contaminated with vismodegib.

You should talk to your study doctor about any side effects that you experience while taking part in the study.

# Risks and side effects related to vismodegib

# Likely (seen in more than 10% of patients)

- Muscle spasms
- Hair loss
- Taste changes, lack of taste function
- Weight loss
- Fatigue or tiredness
- Nausea or the urge to vomit
- Diarrhea
- Loss of appetite
- Constipation
- Vomiting
- Joint aches
- Bloated feeling (dyspepsia)
- Second primary malignancies
- Squamous cell carcinoma
- Abdominal/upper abdominal pain

## Less Likely (seen in 1%-10% of patients)

- Monthly missed periods in females who can become pregnant
- Low levels of sodium in the blood (may cause nausea, lethargy, muscle spasms, or seizures)
- Low potassium levels (may cause irregular heartbeat and breakdown of muscles)
- Higher than normal blood level of urea or other nitrogen-containing compounds in the blood (may cause loss of appetite, lethargy, and mental slowness)
- Lack of energy (asthenia)
- Dehydration
- Pain in extremities
- Loss of eyelashes/eyebrows (madarosis)
- Abnormal hair growth
- Death/sudden death/cardiac death
- Bone fracture
- Venous thromboembolic events
- Fainting (syncope)

ICF 02/22/2017 **PAGE 7 OF 14** CC#122011 Sue S. Yom, MD, and Roy Grekin, MD



- Hepatic enzyme increased
- Blood creatinine phosphokinase increased
- Aspartate aminotransferase increased
- Blood alkaline phosphatase increased
- Pain on one's side between ribs and hip (flank pain)
- Pain in muscles and bones (musculoskeletal pain)
- Back pain
- Muscle pain
- Musculoskeletal chest pain

# Rare (seen in less than 1% of patients)

- Headache
- Confusion
- Liver function test abnormal
- Blood bilirubin increased

## Risks and side effects related to radiation

# <u>Likely</u>

- Sores in the mouth and/or throat which can be painful and make it very difficult to chew and or swallow foods
- Mouth dryness
- Changes in taste and/or smell that may be permanent
- Thick saliva
- Hoarseness
- Tanning or redness and/or irritation of the skin in the head and neck area being treated with radiation
- Ear pain and/or pressure
- Fatique
- Weight loss
- Permanent hair loss in the area treated with radiation
- Loss of teeth, or cavities in the teeth, if strict dental care is not followed and/or hypersensitivity of teeth

# Less Likely, But Serious Effects

- Decrease in function of the thyroid gland that may require you to take thyroid replacement medicine to prevent you from feeling tired or sleepy
- Serious damage to the spinal cord, nerves in the neck, jawbone, voice box, skin, or other
  parts of the head and neck that may require a major operation to correct and, rarely, can
  even be life threatening
- Temporary pain or scarring around nerves in the shoulder that could cause numbness and/or weakness
- Breathing problems
- Difficulty with swallowing and eating for which you might need a long term or permanent feeding tube; possibility of inhaling food and/or liquids into the lungs – which could also result in pneumonia.
- Serious ear infections and/or hearing loss
- Damage to the spinal cord leading to permanent weakness and/or symptoms like a "stroke"
- Permanent hair loss (of the face/chin/neck)

# **Risks related to Study Procedures**

**Surgery and Radiation risk:** If your basal cell carcinoma is advanced, if the disease is left untreated or recurs in the same location after surgery or radiotherapy, it may advance further into surrounding areas such as sensory organs (ears, nose and eyes), bone, or other tissues such as the brain. Depending on the location of the lesion, some cases of advanced BCC can be disfiguring, and treatment with surgery or radiation can lead to the loss of sensory organs and functions such as eyesight or hearing. However these consequences are from the disease or from the surgery/radiation not from vismodegib.

**Study drug combination risks:** The side effects of the combination of vismodegib and radiation are not yet known. Combining vismodegib with radiation to the head and neck can increase the effectiveness of radiation therapy on your cancer, but may increase the side effects of the radiation on normal tissue in the treatment area. You will be monitored closely for side effects and your doctor may change your medications if it appears that this combination is causing serious side effects. You should tell your doctor about any side effects you experience while on this study. When additional information about side effects is known, you will be notified of any further study drug related effects.

**Blood Drawing (venipuncture) risks:** Drawing blood may cause temporary discomfort from the needle stick, bruising, and infection.

**Radiation (X-ray) risks:** As a result of participating in this study, you will receive a significant amount of radiation. The amount is similar to that received in many standard x-ray procedures, but is far more than you would receive from natural daily exposure or in the normal course of treatment, and carries at least a theoretical risk. If you are especially concerned with radiation exposure, you should discuss this with the researchers.

**Chest X-ray risks:** See radiation risks above.

CT scan risks: CT scans involve the risks of radiation (see above). In addition, if contrast material (iodine dye) is used, there is a slight risk of developing an allergic reaction, from mild (itching, rash) to severe (difficulty breathing, shock, or rarely, death). The contrast material may also cause kidney problems, especially if you are dehydrated or have poor kidney function. The study doctors will ask you about any allergies or related conditions before the procedure. If you have any of these problems, you may not be allowed to have a CT scan.

Having a CT scan may mean some added discomfort for you. In particular, you may be bothered by feelings of claustrophobia when placed inside the CT scanner, or by lying in one position for a long time. If contrast material is used, you may feel discomfort when it is injected. You may feel warm and flushed and get a metallic taste in your mouth. Rarely, the contrast material may cause nausea, vomiting or a headache.

**PET/CT scan risks:** The PET/CT scan exposes your body to radiation, see radiation risk above. The radiation levels come from a tracer which is a radioactive chemical injected into a vein in your arm. The tracer lets the doctor see how your cells are functioning and the radiation levels are very low. You may have an allergic reaction to the chemical used in the scan. For some patients, having to lie still on the scanning table for the length of the procedure may cause some discomfort or pain. After the scan your arm may be a little bit sore or have some redness where the IV was placed in your arm. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

**MRI risks:** Because the MRI machine acts like a large magnet, it could move iron-containing objects in the MRI room during your examination, which in the process could possibly harm you. Precautions have been taken to prevent such an event from happening; loose metal objects, like pocket knives or key chains, are not allowed in the MRI room. If you have a piece of metal in your body, such as a fragment in your eye, aneurysm clips, ear implants, spinal nerve

ICF 02/22/2017 PAGE 9 OF 14 CC#122011

stimulators, or a pacemaker, you will not be allowed into the MRI room and cannot have an MRI.

Having an MRI may mean some added discomfort for you. In particular, you may be bothered by feelings of claustrophobia and by the loud banging noise during the study. Temporary hearing loss has been reported from this loud noise. This is why you will be asked to wear ear plugs. At times during the test, you may be asked to not swallow for a while, which can be uncomfortable.

Because the risks to a fetus from MRI are unknown, pregnant women must not participate in this study.

Contrast agent (gadolinium) risks: A few side effects of gadolinium injection such as mild headache, nausea, and local pain may occur. Rarely (less than 1% of the time) low blood pressure and lightheadedness occurs. This can be treated immediately with intravenous fluids. Very rarely (less than one in one thousand), patients are allergic to gadolinium. These effects are most commonly hives and itchy eyes, but more severe reactions have been seen which result in shortness of breath.

Patients with severe kidney disease sometimes have a bad reaction to gadolinium contrast. The condition is called nephrogenic systemic fibrosis (NSF). It can cause skin to tighten or scar and can damage internal organs. Sometimes it can be life-threatening. There are no reports of NSF in patients with normal kidney function. Before you have a MRI scan requiring an injection of gadolinium contrast, you will have a blood test in order to check the function of your kidneys. Based on your medical history and the results of the test, a doctor will decide whether it is safe for you to undergo the MRI scans.

**Tumor biopsy risks:** The general risks associated with this procedure are pain, discomfort, infection, bleeding and injury to organs nearby.

**Reproductive risks:** You should not become pregnant or father a baby while on this study because the drugs in this study can affect an unborn baby.

**Women** should not breastfeed a baby while on this study, or for 24 months after completing therapy. It is important to understand that you need to use birth control while on this study. Women of childbearing age are required to use two forms of acceptable contraception (including one acceptable barrier method with spermicide) during treatment with vismodegib and for 24 months after completing therapy.

**Men** must agree not to donate sperm and are required use condoms at all times, even after a vasectomy, during sexual intercourse with pregnant partners or female partners of childbearing age during treatment with vismodegib and for 3 months after the last dose. Vismodegib is present in semen. It is not known if the amount of vismodegib in semen can cause embryo-fetal harm. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some methods might not be approved for use in this study.

**Unknown Risks:** The experimental treatments may have side effects that no one knows about yet. The researchers will let you know if they learn anything that might make you change your mind about participating in the study.

Blood Donation: Do not donate blood or blood products while on this study and for 24 months after the last dose of vismodegib.

For more information about risks and side effects, ask your study doctor.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

Taking part in this study may or may not make your health better. While doctors hope that vismodegib and radiation will be more useful against your cancer compared to the usual treatment, there is no proof of this. We do know that the information from this study will help doctors learn more about vismodegib and radiationas a treatment for cancer. This information could help future cancer patients.

#### WHAT OTHER CHOICES DO I HAVE IF I DO NOT TAKE PART IN THIS STUDY?

Your other choices may include:

- Getting treatment or care for your cancer without being in a study alternative treatment options such as vismodegib or radiation therapy alone. Both are available off-study.
- Taking part in another study
- Getting comfort care, also called palliative care this type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer; comfort care does not treat the cancer directly, it works to improve how you feel and keep you as active and comfortable as possible
- Getting no treatment

Your physician will discuss these other options with you. Please talk to your doctor about your choices before deciding if you will take part in this study.

# WILL MY MEDICAL INFORMATION BE KEPT PRIVATE?

We will do our best to make sure that the personal information in your medical record is kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- Genentech/Roche Pharmaceuticals and their authorized representatives
- UCSF Committee on Human Research
- The National Cancer Institute (NCI) and other government agencies, e.g., the Food and Drug Administration (FDA), involved in overseeing research
- UCSF Helen Diller Family Comprehensive Cancer Center
- The University of California
- Collaborator sites: Memorial Sloan Kettering

Participation in research may involve a loss of privacy, but information about you will be handled as confidentially as possible. A medical record will be created because of your participation in this study. Your consent form and some of your research test results will be included in this record. Therefore, your other doctors may become aware of your participation. Hospital regulations require that all health care providers treat information in medical records confidentially.

## WHAT ARE THE COSTS OF TAKING PART IN THE STUDY?

You and/or your health plan/insurance company will need to pay for some or all of the costs of treating your cancer in this study. Some health plans will not pay these costs for taking part in studies. Check with your health plan/insurance company to find out what they will pay for. Your study doctors or their clinical staff will obtain authorization from your insurance company prior to beginning your treatment. Taking part in this study may or may not cost you or your insurance company more than the cost of getting regular cancer treatment.

Genentech will supply vismodegib at no charge. Additionally, you will not be billed for research

IRB NUMBER: 13-10524 IRB APPROVAL DATE: 02/08/2018

IRB EXPIRATION DATE: 02/07/2019

procedures required specifically by the study. Research procedures are the Skindex-16 survey and digital photographs. Other procedures, which are also done in this study but are part of your normal care, will be paid for by you or your insurance. This includes radiation therapy and physical exams that are considered part of the standard treatment for your cancer. You or your insurance company will be billed for the radiation therapy.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at http://cancer.gov/clinicaltrials/understanding/insurance-coverage. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

#### WILL I BE PAID FOR TAKING PART IN THIS STUDY?

You will not be paid for taking part in this study.

## WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THIS STUDY?

It is important that you tell your study doctor Sue S. Yom, MD or Roy Grekin, MD if you feel that you have been injured because of taking part in this study. You can tell her in person or call her

Treatment and Compensation for Injury: If you are injured as a result of being in this study, the University of California will provide necessary medical treatment. The costs of the treatment may be billed to you or your insurer just like any other medical costs, or covered by the University of California or Genentech, depending on a number of factors. The University and the study sponsor do not normally provide any other form of compensation for injury. For further information about this, you may call the office of the Committee on Human Research at 415-476-1814.

#### WHAT ARE MY RIGHTS IF I TAKE PART IN THIS STUDY?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

### WHO CAN ANSWER MY QUESTIONS ABOUT THE STUDY?

You can talk to your study doctor about any questions, concerns, or complaints you have about this study. Contact your study doctor Sue S. Yom MD or Roy Grekin

If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you may have about the study, please call the Office of the Committee on Human Research at 415-476-1814

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



# **CONSENT**

You have been given copies of this consent form and the Experimental Subject's Bill of Rights to keep.

You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to participate or to withdraw at any point in this study without penalty or loss of benefits to which you are otherwise entitled.

If you wish to participate in this study, you should sign below.

Witness – Only required if the participant is a non-English speaker

Participant Date

Participant name (print)

Person obtaining consent Date

Person obtaining consent (print)

Date

#### Prohibited Medications and Foods to Avoid

During your participation in this study you will not be able to take certain medications. The following tables provide a list of <u>prohibited</u> medications and a list of medications to avoid while you are on this study. If you go to any medical visit, please take this list with you for the doctor's reference. If you need to take any of the medications on the list during the study, you will be able to, but you may be removed from the study.

Before you begin treatment, Dr. Yom or one of her associates will review all medications you are taking. Make sure you talk with Dr. Yom before you start or stop taking any medications. This list contains only the most common drugs and food that are known to interact with the drugs used in this study. It is very important to discuss all medications that you are taking with your study doctor. This information will be reviewed at each study visit.

In addition to the listed medications, you should also avoid eating grapefruit and grapefruit juices.

| | <u>2C9</u> | <u>2C19</u> |
|---|---|---|
| <u>Miscellaneous</u> : | <u>NSAIDs</u> : | Proton Pump Inhibitors: |
| repaglinide | Diclofenac | omeprazole |
| rosiglitazone | Ibuprofen | lansoprazole |
| | piroxicam | pantoprazole |
| | naproxen | rabeprazole |
| | celecoxib | esoprazole |
| | Oral Hypoglycemic Agents: | Anti-epileptics:<br>diazepam |
| | glipizide | phenytoin |
| | tolbutamide | phenobarbitone |
| | | • |
| | Angiotensin II Blockers: | Miscellaneous: |
| | | amitriptyline |
| | irbesartan | clomipramine |
| | losartan | clopidogrel |
| | NOT candesartan | cyclophosphamid<br>e progesterone |
| | NOT valsartan | o progessione |
| | Miscellaneous: | |
| | fluvastatin | |
| | phenytoin | |
| | sulfamethoxazole | |
| | tamoxifen torsemide | |
| | warfarin | |